CLINICAL TRIAL: NCT04509583
Title: Is Micro Nutrient Supplement Effective in Improving the Sperm DNA Fragmentation
Brief Title: The Role of Micro Nutrient Supplement in Improvement of the Sperm DNA Fragmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hue University of Medicine and Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H2019/433
Record Dates: First submitted 2020-05-05; First posted 2020-08-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-02

CONDITIONS: Infertility, Male
Keywords: Sperm DNA fragmentation; micronutrient; In vitro fertilization
MeSH Terms: conditions — Infertility, Male | interventions — Vitamin E

STUDY DESIGN:
Intervention Model Description: Men from infertile couples with increased sperm DNA fragmentation will be randomized devided into 2 groups: (1) with multi-micronutrient supplements (PROFortilTM) plus Vitamin E and (2) with Vitamin E only.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Computerized label randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PROFortil group (Experimental): Men with increased sperm DNA fragmentation (>=30%) will be indicated for multi-micronutrient supplement (PROfortil™, twice daily) plus Vitamin E (Enat 400, once per day) in 3 months then checked again post-treatment for DF).
  The IVF/ICSI cycles will then be analyzed for embryo quality, pregnancy outcomes including biochemical pregnancy rate, clinical pregnancy rate, on-going pregnancy, miscarriage.
  Interventions: Dietary Supplement: PROFortil
- Vitamin E group (Other): Any case with high DNA fragmentation index (DFI >=30%) will be randomized indicated only Vitamin E (Enat 400 once per day) in 3 months then checked again post-treatment for (DFI).
  The IVF/ICSI cycles will then be analyzed for embryo quality, pregnancy outcomes including biochemical pregnancy rate, clinical pregnancy rate, on-going pregnancy, miscarriage.
  Interventions: Other: Vitamin E

INTERVENTIONS:
Dietary Supplement: PROFortil — Multi-micronutrient supplement (PROfortil™, twice daily) plus Vitamin E (Enat 400, once per day) in 3 months
  Arms: PROFortil group
Other: Vitamin E — Only Vitamin E (Enat 400, once per day) in 3 months
  Arms: Vitamin E group

SUMMARY:
Male from infertile couples are tested for semen analysis and sperm DNA fragmentation. Any case with high DNA fragmentation index (DFI) will be randomized indicated for multi-micro nutrient supplement (PROfortil™) in 3 months and then checked again post-treatment for (DFI). The IVF/ICSI cycles will be analyzed for pregnancy outcomes

DETAILED DESCRIPTION:
Higher DFI is correlated with poor embryo development, lower implantation rate in intracytoplasmic sperm injection (ICSI) cycles and higher miscarriage rate.

The effectiveness of micro nutrients (PROfortil™) has been proven in improving sperm quality including sperm cell density, progressive motility and normal morphology.

This randomized controlled trial includes male from infertile couples treated at the Center for Reproductive Endocrinology and Infertility, Hue University hospital, Vietnam from November 2019 to November 2020.

The semen samples were collected from the husband after 3-5 days of abstinence and then evaluated for sperm motility, vitality, concentration and morphology by the guideline of World Health Organization (WHO) 2010.

Sperm DNA fragmentation (SDF) was measured using a sperm chromatin dispersion (SCD) test (Halosperm® kit, Halotech, Madrid, Spain). A total of 500 sperms were examined by only one highly trained technician to decrease variability. DFI was expressed as the percentage of sperms with small halo, without halo and degraded sperms over total of 500 sperms.

Any case with high DNA fragmentation index (DFI >=30%) will be randomized indicated for (group 1) micro nutrient supplement (PROfortil™, twice daily) plus Vitamin E (Enat 400, once per day) in 3 months and (group 2) only Vitamin E (Enat 400 once per day) then checked again post-treatment for (DFI).

The IVF/ICSI cycles will then be analyzed for embryo quality, pregnancy outcomes including biochemical pregnancy rate, clinical pregnancy rate, on-going pregnancy, miscarriage.

ELIGIBILITY:
Inclusion Criteria:

- Male from infertile couples

Exclusion Criteria:

* Men with acute systemic diseases
* acute urinary tract infection
* hepatic function disorders
* malignant diseases
* retrograde ejaculation
* azoospermia

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
The change of DFI after micro nutrients supplements | 3 months
  The change of sperm DNA Fragmentation Index after treatment with PROfortil in 3 months

SECONDARY OUTCOMES:
The impact of micro nutrients supplements on embryo quality after ICSI | 3 months
  The blastocyst quality in IVF/ICSI cycles after treatment with PROFortil
The impact of micro nutrients supplements on pregnancy outcomes after ICSI | 3 months
  The pregnancy rate in IVF/ICSI cycles after treatment with PROFortil

CONTACTS AND LOCATIONS:
Overall Officials: Minh Tam Le, M.D.,Ph.D, Study Director — Hue University of Medicine and Pharmacy, Hue University
Locations (1):
- Hue University of Medicine and Pharmacy, Hue University, Huế, Thua Thien, Vietnam

REFERENCES:
- [Derived] Nguyen ND, Le MT, Tran NQT, Nguyen QHV, Cao TN. Micronutrient supplements as antioxidants in improving sperm quality and reducing DNA fragmentation. Basic Clin Androl. 2023 Sep 14;33(1):23. doi: 10.1186/s12610-023-00197-9. PMID 37704942